CLINICAL TRIAL: NCT06579495
Title: Effects of Competitive Exergame on Weight Loss, Mental Health, and Social-emotional Among Overweight and Obese Male Adolescents in China
Brief Title: Effects of Competitive Exergame on Weight Loss, Mental Health, and Social-emotional
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Liu Chunqing, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Liu Chunqing
Record Dates: First submitted 2024-08-25; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Weight Loss; Mental Health Issue; Overweight and Obesity
Keywords: Competitive Exergame; Mental Health; Social-emotional
MeSH Terms: conditions — Weight Loss; Overweight; Obesity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: In this experiment, experimental group 1 involved peer participation in a Competitive Exergame; that is, the participants were accompanied by peers to complete the experiment. Experimental group 2 completed the task on their own using the Single-player Competitive Exergame. The control group did not undergo any intervention and simply continued with their normal school routine.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer involvement in Two player mode(peer involvement) in Competitive Exergame play (Experimental): The peer participation group requires a classmate to accompany the child to complete the experiment task.
  Interventions: Other: Peer involvement in Two player mode(peer involvement) in Competitive Exergame play
- Single player mode in Competitive Exergame play (Experimental): Single player mode play the single-person model and the child need to complete the experimental task under the teacher's supervision.
  Interventions: Other: Single player mode in Competitive Exergame play
- Children did not engage in any Competitive Exergame play (Active Comparator): Children did not engage in any Competitive Exergame play nor any other structured school-based PA programs beyond physical education, and maintained just for a normal school life.
  Interventions: Other: Children did not engage in any Competitive Exergame play

INTERVENTIONS:
Other: Peer involvement in Two player mode(peer involvement) in Competitive Exergame play — Device: Nintendo Wii sports competitive versus. The duration of the study was 8 weeks and the frequency was 45 minutes, three times per week. In the first two weeks, three games of bowling, tennis and fencing will be selected for experimentation at the beginner and intermediate levels respectively. In the three weeks from week 3 to week 5, golf, tennis and cycling were selected for the beginner, intermediate and advanced levels of the experiment. In the last three weeks, basketball, boxing and dancing will be selected for experimentation at beginner, intermediate and advanced levels respectively. The control group did not participate in any intervention and maintained daily physical activity behavior.
  Arms: Peer involvement in Two player mode(peer involvement) in Competitive Exergame play
Other: Single player mode in Competitive Exergame play — Device: Nintendo Wii sports competitive versus. The duration of the study was 8 weeks and the frequency was 45 minutes, three times per week. In the first two weeks, three games of bowling, tennis and fencing will be selected for experimentation at the beginner and intermediate levels respectively. In the three weeks from week 3 to week 5, golf, tennis and cycling were selected for the beginner, intermediate and advanced levels of the experiment. In the last three weeks, basketball, boxing and dancing will be selected for experimentation at beginner, intermediate and advanced levels respectively. The control group did not participate in any intervention and maintained daily physical activity behavior.
  Arms: Single player mode in Competitive Exergame play
Other: Children did not engage in any Competitive Exergame play — Device: Nintendo Wii sports competitive versus. The duration of the study was 8 weeks and the frequency was 45 minutes, three times per week. In the first two weeks, three games of bowling, tennis and fencing will be selected for experimentation at the beginner and intermediate levels respectively. In the three weeks from week 3 to week 5, golf, tennis and cycling were selected for the beginner, intermediate and advanced levels of the experiment. In the last three weeks, basketball, boxing and dancing will be selected for experimentation at beginner, intermediate and advanced levels respectively. The control group did not participate in any intervention and maintained daily physical activity behavior.
  Arms: Children did not engage in any Competitive Exergame play

SUMMARY:
Overweight and obesity are prevalent, especially among adolescents. By 2016, over 124 million children and adolescents, comprising 6% of girls and 8% of boys, were classified as obese. Over the past century, childhood obesity has transitioned from a symbol of prosperity and well-being to being acknowledged as a significant health concern. Furthermore, according to the World Health Organization, it is now considered "one of the most serious challenges of the 21st century." Overweight and obese adolescents have serious problems with weight loss, mental health and social-emotional. A previous study by Lopez identified time constraints and a lack of motivation as hindrances to physical activity, a key component of effective weight loss measures.

In today's society, developed modern technology plays a very important role in the growth of teenagers and in their daily life. Exergame is a new type of video game that allows participants to be more active, stimulating their whole body movement game experience and promoting non-sedentary physical activity. Active Video Games (AVGs) utilize motion-sensing technology to simplify the complex functions typically associated with computer operations. Exergaming is a novel video game that stimulates an active whole-body gaming experience that allow to play multiple players compete or cooperate on a team. Playing against a peer offering both virtual and real social interaction is more likely to sustain engagement, and also promotes higher energy expenditure in an exergame compared to playing alone.

Harnessing adolescents' fascination with video games represents an innovative strategy in the battle against pediatric obesity and sedentary lifestyles. It is especially important to intervene with overweight and obese adolescents using Competitive exergame to become more actively involved in sports, no longer afraid of social interaction, and improve quality of life. Competitive exergame provides a virtual and a real social interaction to improve mental health on overweight and obese adolescents. Therefore, the study will systematically investigate the effects of Competitive Exergame on Weight loss, Mental health,and Social-emotional among overweight and obese male adolescents in China.

DETAILED DESCRIPTION:
To assess the effectiveness of Competitive exergame as an intervention, overweight and obese adolescents participating in this study were randomly assigned to three groups (two experimental and one control). This experimental design consists of peer involvement in AVG play and AVG single-player, as well as one control group (children maintained normal daily life without intervention). The sample is 12-14-year-old Chinese overweight and obese male middle school students. The test site is in the school, and the child needs to complete the experimental task under the PE teacher's supervision. The researchers will set up their groups on the WeChat platform, which will be used to contact parents to learn about the subjects' daily diets. The experiment lasted for 8 weeks, with the experimental group conducted three 45-minute interventions per week. The independent variable in this study was the Competitive Exergame intervention, while the dependent variables were weight loss, mental health, and social-emotional. Based on the study design, which involves learning from and summarizing quantitative studies, the dependent variables were measured at three points: pre-test (before the intervention), post-test 1 (4 weeks after the intervention), and post-test 2 (8 weeks after the intervention). The data from these three measurements were collected, organized, and analyzed.

BMI was calculated using a formula, body fat was measured using bioelectrical impedance (BIA), and waist-to-hip ratio was measured using an accurate tape measure. Satisfaction was measured using Multidimensional Students' Life Satisfaction Scale (MSLSS). It should be noted that a 6-point agreement format has been used with middle and high school students. For each item, there are 4 response options ranging from 1 to 6 (1=Strongly Disagree'2=Mostly Disagree, 3=Mildly Disagree'4=Mildly Agree'5=Mostly Agree'6=Strongly Agree). Hence'10 negatively-keyed items are scored so that Strongly Agree= 1, and so forth. Higher scores thus indicate higher levels of life satisfaction throughout the scale. Previous studies have confirmed the Cronbach's alpha is 0.90. Self-confident was measured using Self-Confidence Scale for Chinese Primary and Secondary School (SCS). A 17-item self-confidence scale for primary and secondary school students in China was developed through theoretical construction exploratory and confirmatory factor analysis. The SCS used a 5-point Likert scale ranging from 1 (disagree a lot) to 5 (agree a lot). A higher score indicates a student perceived higher Self-Confidence. The scale has been validated with a Cronbach's alpha of 0.84. Depression was measured using Patient Health Questionnaire (PHQ-9). It comprises 9 diagnostic symptom criteria based on the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) major depressive disorder. Each item has 4 response options ranging from 0 = "not at all" to 3 ="nearly every day" with total scores ranging from 0 to 27. Previous studies have confirmed the Cronbach's alpha is 0.89. Self-efficacy was measured using Physical activity self-efficacy Scales (S-PASESC). The SPASES used a 5-point Likert scale ranging from 1 (disagree a lot) to 5 (agree a lot). A higher score indicates a student perceived higher PA self-efficacy. A higher score indicates a student perceived higher PA self-efficacy. The scale has been validated with a Cronbach's alpha of 0.92. Self-esteem was measured using Self-Esteem Scale (SES). A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. All items are answered using a 4-point Likert scale ranging from strongly agree to strongly disagree. Items 2, 5, 6, 8, 9 are reverse scored. Give "Strongly Disagree" 1 point, "Disagree" 2 points, "Agree" 3 points, and "Strongly Agree" 4 points. The scores for all ten items. Keep scores on a continuous scale. Higher scores indicate higher self-esteem. The scale has been validated with a Cronbach's alpha of 0.88. Social Anxiety was measured using Social Phobia and Anxiety Inventory Form (SPAI-B). The SPAI-B consists of 16 items answered with a 5-point Likert scale ranging from 1 (Never happens) to 5 (Always happens). The total score is 23 to 115, and the higher the score, the more obvious the anxiety symptoms. The scale has been validated with a Cronbach's alpha of 0.92.

Before the training was conducted, training and explanations were provided to all members of the experimental group, which mainly included game mode selection, game login, and explanation of operating procedures. The game consists of 9 sports events. Each game has a single-player mode and a multi-player mode. Each class consists of three parts: Upper and lower body training, Sports games and Aerobic exercise. Players need to choose the mode to exercise. The experiment lasted for 8 weeks, with 45-minute intervention three times a week.

Week 1: Log in to the Nintendo game account registered in advance. Experimental group 1 chose the multiplayer mode and the Experimental group 2 chose the single mode. Each class of Upper and lower body strength training (Bowling) section lasts 10 minutes. The Sports games (Table tennis) section of each lesson lasts 20 minutes, and the Cardio (Fecing) section of each lesson lasts 15 minutes. This week's game level is Beginner.

Week 2: Following the game selections from last week, there is a multiplayer mode for Experimental Group 1 and a single-player mode for Experimental Group 2. This week's game level is Advanced.

Week 3: Experimental group 1 chose the multiplayer mode and the Experimental group 2 chose the single mode. Each class of Upper and lower body strength training (Golf) section lasts 10 minutes. The Sports games (Tennis) section of each lesson lasts 20 minutes, and the Cardio (Cycling) section of each lesson lasts 15 minutes. This week's game level is Beginner.

Week 4: Following the game selections from last week, there is a multiplayer mode for Experimental Group 1 and a single-player mode for Experimental Group 2. This week's game level is Intermediate.

Week 5: Following the game selections from last week, there is a multiplayer mode for Experimental Group 1 and a single-player mode for Experimental Group 2. This week's game level is Advanced.

Week 6: Experimental group 1 chose the multiplayer mode and the Experimental group 2 chose the single mode. Each class of Upper and lower body strength training (Basketball) section lasts 10 minutes. The Sports games (Boxing) section of each lesson lasts 20 minutes, and the Cardio (Dance) section of each lesson lasts 15 minutes. This week's game level is Beginner.

Week 7: Following the game selections from last week, there is a multiplayer mode for Experimental Group 1 and a single-player mode for Experimental Group 2. This week's game level is Intermediate.

Week 8: Following the game selections from last week, there is a multiplayer mode for Experimental Group 1 and a single-player mode for Experimental Group 2. This week's game level is Advanced.

ELIGIBILITY:
Inclusion Criteria:

* The age of the experimental subjects should be 12-14 years old;
* The student had never played AVG before;
* The students' BMI percentile should be more than 85;
* There are no other sports besides daily physical activities;
* The students without physical and/or mental disabilities;

Exclusion Criteria:

* Having self-reported physical and/or mental disabilities;
* Having motion sickness reaction when exercising under AVG based condition;
* Relevant weight loss medicine taken within half a year;

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Weight | pretest, week 4, week 8
  Weight is measured using a standard kilogram scale and results are given in kilograms (kg).
Height | pretest, week 4, week 8
  Height is measured using a standard height ruler and results are given in meters(m).
Body Mass Index (BMI) | pretest, week 4, week 8
  Body Mass Index (BMI) is measured using the formula BMI = weight (kg)/height (m)^2.
Waist-to-hip ratio | pretest, week 4, week 8
  Waist-to-hip ratio is measured using a precise tape measure, with waist and hip measurements expressed in centimeters (cm).
Body fat | pretest, week 4, week 8
  Body fat was measured by a body composition analyzer using bioelectric impedance analysis (BIA), and the results were expressed in %.
The Multidimensional Students' Life Satisfaction Scale (MSLSS) | pretest, week 4, week 8
  The Multidimensional Students' Life Satisfaction Scale (MSLSS) is designed to provide a profile of children's life satisfaction across key domains. It should be noted that a 6-point agreement format has been used with middle and high school students. Higher scores thus indicate higher levels of life satisfaction throughout the scale.
Self-Confidence Scale for Chinese Primary and Secondary School (SCS) | pretest, week 4, week 8
  Self-confidence was measured using Self-Confidence Scale for Chinese Primary and Secondary School (SCS). The SCS used a 5-point Likert scale ranging from 1 (disagree a lot) to 5 (agree a lot). A higher score indicates a student perceived higher Self-Confidence.
Patient Health Questionnaire (PHQ-9) | pretest, week 4, week 8
  A higher score indicates a student perceived higher. Self-Confidence. Depression wsa measured using Patient Health Questionnaire (PHQ-9). It comprises 9 diagnostic symptom criteria based on the Diagnostic and Statistical Manual of Mental Disorders#IV (DSM#IV) major depressive disorder.
Physical activity self-efficacy Scales (S-PASESC) | pretest, week 4, week 8
  Self-efficacy was measured using Physical activity self-efficacy Scales (S-PASESC). The SPASES used a 5-point Likert scale ranging from 1 (disagree a lot) to 5 (agree a lot). A higher score indicates a student perceived higher PA self-efficacy. A higher score indicates a student perceived higher PA self-efficacy.
Self-Esteem Scale (SES) | pretest, week 4, week 8
  Self-Esteem was measured uasing Self-Esteem Scale (SES). A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. All items are answered using a 4-point Likert scale ranging from strongly agree to strongly disagree. The scores for all ten items. Keep scores on a continuous scale. Higher scores indicate higher self-esteem.
Social Phobia and Anxiety Inventory Form (SPAI-B) | pretest, week 4, week 8
  Social Anxiety was measured using Social Phobia and Anxiety Inventory Form (SPAI-B). The SPAI-B consists of 16 items answered with a 5-point Likert scale ranging from 1 (Never happens) to 5 (Always happens). The total score is 23 to 115, and the higher the score, the more obvious the anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Chunqing Liu, Principal Investigator — Universiti Putra Malaysia

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I don't want to share it until after graduation.

REFERENCES:
- [Result] Irandoust K, Taheri M, H'mida C, Neto GR, Trabelsi K, Ammar A, Souissi N, Chtourou H, Nikolaidis PT, Rosemann T, Knechtle B. Exergaming and Aquatic Exercises Affect Lung Function and Weight Loss in Obese Children. Int J Sports Med. 2021 Jun;42(6):566-572. doi: 10.1055/a-1289-9307. Epub 2020 Nov 11. PMID 33176381
- [Result] Christison AL, Evans TA, Bleess BB, Wang H, Aldag JC, Binns HJ. Exergaming for Health: A Randomized Study of Community-Based Exergaming Curriculum in Pediatric Weight Management. Games Health J. 2016 Dec;5(6):413-421. doi: 10.1089/g4h.2015.0097. Epub 2016 Dec 2. PMID 27911621